CLINICAL TRIAL: NCT06414746
Title: A Multicenter Observational Retrospective-prospective Study of Prevalence, Clinical Characteristics of Hereditary Transthyretin Amyloidosis Polyneuropathy in Russian Patients Undergoing Surgery for CTS in Real Clinical Practice
Brief Title: Hereditary Transthyretin Amyloidosis Polyneuropathy in Patients With Carpal Tunnel Syndrome in Russia
Acronym: LOCUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8451R00001
Record Dates: First submitted 2024-02-16; First posted 2024-05-16 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Transthyretin Amyloidosis; Carpal Tunnel Syndrome; Polyneuropathy; Amyloidosis
Keywords: ATTR PN; CTS; PN; carpal tunnel syndrome; polyneuropathy; amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Carpal Tunnel Syndrome; Polyneuropathies; Amyloidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter observational study consisting of retrospective and prospective phases. The retrospective phase will entail secondary data collection from electronic or paper medical records of patients who underwent surgery for CTS to assess their probability of having ATTR PN.

DETAILED DESCRIPTION:
ATTR PN is a genotypically, phenotypically and geographically variable disease with a poor prognosis, albeit available disease-modifying drugs can change the disease trajectory. Thus country-specific epidemiologic data collection and identification of early stage PN, including previously misdiagnosed patients, is crucial to improve outcomes and quality of life. However, no observational studies on the epidemiology of ATTR PN in the whole Russian population, or in patients with CTS, have been performed.

Therefore, there is a need to conduct a large-scale observational study to determine the prevalence of ATTR PN in Russia, obtain information on patients' clinical characteristics, and determine their medical needs.

The approaches to diagnosis of ATTR PN in Russia over the past few years have been characterized by the use of heterogenous methods, partially explained by the lack of availability of molecular genetic testing, which is essential to diagnose the presence of pathogenic mutation in patients with hereditary ATTR PN. Thus, recent introduction of such tests into routine clinical practice may allow to assess reliable epidemiologic data including estimation of true ATTR PN prevalence among patients with CTS, which can often be the first manifestation of the disease. Earlier recognition, in turn, may lead to timely treatment initiation and change in the prognostic outlook of ATTR PN patients.

In order to assess the prevalence of ATTR PN in patients undergoing surgery for CTS in Russia this study will retrospectively include patients with the diagnosis of CTS undergoing surgery between the 1st January 2021 and the 1st September 2024. Suspicion of ATTR PN will be assessed in each case, and diagnostic tests (comprehensive neurological examination including nerve conduction study (NCS) combined with molecular genetic testing) to confirm or exclude the disease will be conducted prospectively in eligible patients. In addition to that, clinical features, concomitant manifestations, and diagnosed genotypes will be analyzed to examine characteristic ATTR PN patient profiles in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

for the retrospective phase are:

1. Patients with the established diagnosis of CTS.
2. Bilateral involvement of carpal tunnel established between the 1st January 2021 and the 31st December 2024 (both patients who underwent CTS surgical intervention and without it are enrolled).
3. Age ≥ 18 years at the time of CTS diagnosis.
4. Provided written informed consent for the prospective phase of the study (including molecular genetic testing).
5. Presence of ≥1 of the following features (red flags):

   a. CIDP or polyneuropathy of unknown etiology in the family history; b. Spinal canal stenosis of the lumbar region; c. Autonomic dysfunction, defined by the presence of ≥1 of the following symptoms - i. Gastrointestinal complaints (constipation, chronic diarrhea, or both); ii. Erectile dysfunction; iii. Orthostatic hypotension; d. Gait disorders; e. Sweating disorders, anhidrosis. f. Paresthesia and burning of the skin of the distal extremities g. Distal symmetrical paresis h. Hypotrophy and hypotension of limb muscles, areflexia i. Biceps tendon rupture j. Aortic valve stenosis k. Diagnosis of HFpEF

   l. Unexplained weight loss ≥5 kilos at any timepoint since the onset of symptoms of CTS; m. Left ventricular hypertrophy (based on electro- or echocardiographic criteria documented in the patient's medical record); n. Heart rhythm disorders; o. Renal abnormalities, defined by ≥1 of the following features - i. Documented diagnosis of chronic kidney disease (CKD); ii. Decreased estimated glomerular filtration rate (eGFR <60 mL/min/1.73m2); iii. Increased serum creatinine (SCr) above reference range of the local laboratory; iv. Albuminuria (≥30 mg/g of creatinine or ≥30 mg/24h); v. Proteinuria (according to urinalysis results); p. Ophthalmology disorder defined by ≥1 of the following features - i. Vitreous body inclusions (opacification); ii. Glaucoma; iii. Pupillary disorders; iv. Vitrectomy
6. Absence of previously established ATTR PN diagnosis (ICD-10 code Е85.1, "Neuropathic hereditary familial amyloidosis").

Exclusion Criteria:

1. Participation in any interventional trial within the period since identification of bilateral involvement of carpal tunnel until the end of current study.

   The following criteria apply for non-inclusion of patients into the prospective part of the study:
2. Previously performed TTR genetic testing;
3. Verified B12 deficiency;
4. History of alcohol abuse according to the patient's medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter observational study will retrospectively include 1300 consecutive adult patients diagnosed with CTS and having bilateral involvement in Russia from the earliest date of diagnosis to a later one within the specified time period who are observed and monitored at 20 participating sites, including approximately ~800 patients with CTS and high suspicion of having ATTR PN who will be enrolled in the prospective phase.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
To define the prevalence of ATTR PN in patients diagnosed with CTS and having bilateral involvement in routine clinical practice in the Russian Federation. | Up to 12 months
  In order to achieve primary objective, the proportion of patients with confirmed diagnosis of ATTR PN (presence of TTR gene mutation according to the results of molecular genetic testing and clinical symptoms and/or signs of polyneuropathy) among those diagnosed with CTS and having bilateral involvement will be calculated.

SECONDARY OUTCOMES:
To assess general demographic characteristics of patients with ATTR PN in Russia - Mean age (years) at the onset of CTS symptoms | up to 12 months
To assess general demographic characteristics of patients with ATTR PN in Russia: Mean age (years) at the onset of polyneuropathy symptoms | up to 12 months
to assess general demographic characteristics of patients with ATTR PN in Russia: Proportion of patients with late (>50 years) diagnosis of ATTR PN | up to 12 months
to assess general demographic characteristics of patients with ATTR PN in Russia: Mean age (years) at the time of CTS surgery | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia - Number and proportion of patients with specific characteristics of the first and repeat CTS surgery | up to 12 months
  1. Left hand;
  2. Right hand;
  3. Both hands;
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Proportion of patients with CTS recurrence after surgery | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Proportion of patients undergoing repeat surgery for CTS after the index operation | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Proportion of patients with PN progression after surgery | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia - Proportion of patients with different number of red flags: | up to 12 months
  1. 1 red flag;
  2. 2 red flags;
  3. 3 red flags;
  4. 4-5 red flags;
  5. 6-10 red flags;
  6. >10 red flags;
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Mean age (years) at ATTR PN diagnosis | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Proportion of women and men | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia - Mean body mass index (BMI) and proportion of patients with different BMI dimensions at the time of CTS diagnosis and at Visit 1: | up to 12 months
  1. Underweight (BMI <18.5 kg/m2);
  2. Normal weight (BMI ≥18.5 and <25 kg/m2);
  3. Overweight (BMI ≥25 and <30 kg/m2);
  4. Obesity (BMI ≥30 kg/m2)
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Proportion of patients with a history of unexplained weight loss (≥5 kg) at any point since CTS diagnosis | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Mean and median time from CTS symptom onset (months) to ATTR PN diagnosis | up to 12 months
To assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Median number of physicians seen since symptom onset before the correct ATTR PN diagnosis | up to 12 months
To assess general demographic and clinical characteristics of patients with ATTR PN in Russia: Median number of hospitalizations for PN before the correct ATTR PN diagnosis | up to 12 months
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia - Number and proportion of patients with previously established incorrect diagnosis according to medical records, specifically with: | up to 12 months
  1. CIDP;
  2. Lumbar/sacral radiculopathy;
  3. Lumbar canal stenosis;
  4. Paraproteinaemic peripheral neuropathy;
  5. Chronic progressive sensory/sensorimotor axonal idiopathic PN;
  6. AL amyloidosis;
  7. Fibromyalgia;
  8. Other (specify)
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN: Proportion of patients with family history of neuropathic disease | up to 12 months
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN: Proportion of patients with specific peripheral neurological manifestations: | up to 12 months
  1. Neuropathic pain (allodynia, hyperalgesia);
  2. Progressive sensory disturbances (loss of temperature, pain, other sensation);
  3. Paresthesia, dysesthesia;
  4. Progressive motor disturbances;
  5. Walking difficulty, gait disorder;
  6. Balance disorder
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN: Proportion of patients with specific Polyneuropathy Disability (PND) classes: | up to 12 months
  1. 0;
  2. I;
  3. II;
  4. IIIA;
  5. IIIB;
  6. IV;
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - Proportion of patients with specific distribution of polyneuropathy symptoms: | up to 12 months
  1. Upper-limb;
  2. Lower-limb;
  3. Both upper-limb and lower-limb
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - Number of patients with autonomic neurological manifestations, including specifically: | up to 12 months
  1. Orthostatic hypotension;
  2. Syncope;
  3. Gastrointestinal motility disorders - i. Constipation; ii. Early satiety; iii. Diarrhea; iv. Nausea, vomiting;
  4. Erectile dysfunction;
  5. Neurogenic bladder;
  6. Recurrent urinary infections;
  7. Anhidrosis;
To describe data on the presence of cardiovascular, neurological and other comorbidities- Number and proportion of patients taking specific groups of cardiovascular medications at the time of CTS diagnosis and at the time of prospective visit: | up to 12 months
  1. Left ventricular hypertrophy;
  2. Left bundle branch block;
  3. Atrioventricular block;
  4. Heart failure with preserved ejection fraction;
  5. Elevated serum N-terminal-proB-type natriuretic peptide (NT-proBNP) concentration;
  6. Cardiac valve stenosis;
  7. Cardiac valve regurgitation;
  8. Tachyarrhythmia;
  9. Other (specify);
  10. None;
Number of patients taking specific groups of cardiovascular medications at the time of CTS surgery and at the time of prospective visit: | up to 12 months
  1. Angiotensin converting enzyme inhibitor (ACEI) (specify);
  2. Angiotensin receptor blocker (ARB) (specify);
  3. Angiotensin receptor and neprilysin inhibitor (ARNI);
  4. Sodium-glucose transporter type 2 inhibitor (SGLT2i) (specify);
  5. Mineralocorticoid receptor antagonist (MRA) (specify);
  6. Beta-blocker (specify);
  7. Diuretic (specify);
  8. Other cardiovascular (CV) medications (specify);
  9. Other (specify);
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - Number of patients with concomitant ophthalmologic manifestations, including specifically | up to 12 months
  1. Vitreous body inclusions (opacification);
  2. Glaucoma;
  3. Abnormal conjunctival vessels;
  4. Papillary abnormalities;
  5. Dry eye;
  6. Other (specify);
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - Number of patients with concomitant musculoskeletal manifestations, including specifically: | up to 12 months
  1. Spinal stenosis;
  2. Osteoarthritis, including hip and knee arthroplasty;
  3. Trigger finger;
  4. Charcot's joints;
  5. Biceps tendon rupture;
  6. Rotator cuff injury;
  7. Other (specify);
Mean and median serum NT-proBNP (pg/ml) concentration | up to 12 months
Proportion of patients with laboratory confirmed paraproteinemia | up to 12 months
Mean and median urine albumin-creatinine ratio (UACR, mg/g of creatinine) | up to 12 months
Proportion of patients with diagnosed CKD, including specifically | up to 12 months
  1. Stage C1;
  2. Stage C2;
  3. Stage C3a;
  4. Stage C3b;
  5. Stage C4;
  6. Stage C5;
Number of patients with concomitant renal dysfunction, including specifically | up to 12 months
  1. Elevated SCr level (based on the local laboratory reference range);
  2. Decreased eGFR (<60 ml/min/1.73m2);
  3. Presence of albuminuria (≥30 mg/g creatinine (≥30 mg/g of creatinine or ≥30 mg/24h);
  4. Presence of proteinuria (according to urinalysis results);
  5. Ultrasound signs of amyloid nephropathy;
Number of patients with confirmed length-dependent peripheral sensory-motor neuropathy based on NCS results | up to 12 months
Mean and median measured peripheral sensory nerve conduction velocities | up to 12 months
  1. Left Medial;
  2. Left Ulnar;
  3. Left Sural;
  4. Right Medial;
  5. Right Ulnar;
  6. Right Sural;
Number of patients with reduced peripheral sensory nerve conduction velocity at ≥1 site | up to 12 months
Mean and median measured peripheral motor nerve conduction velocities | up to 12 months
  1. Left Medial;
  2. Left Ulnar;
  3. Left Tibial;
  4. Left Peroneal;
  5. Right Medial;
  6. Right Ulnar;
  7. Right Tibial;
  8. Right Peroneal;
Number of patients with reduced motor sensory nerve conduction velocity at ≥1 site | up to 12 months
Mean and median measured sensory action potential (SAP) amplitudes | up to 12 months
  1. Left Medial;
  2. Left Ulnar;
  3. Left Sural;
  4. Right Medial;
  5. Right Ulnar;
  6. Right Sural
Number of patients with reduced/absent SAP amplitude at ≥1 site | up to 12 months
Mean and median measured distal compound muscle action potential (dCMAP) amplitudes | up to 12 months
  1. Left Medial;
  2. Left Ulnar;
  3. Left Tibial;
  4. Left Peroneal;
  5. Right Medial;
  6. Right Ulnar;
  7. Right Tibial;
  8. Right Peroneal
Mean and median measured proximal compound muscle action potential (pCMAP) amplitudes | up to 12 months
  1. Left Medial;
  2. Left Ulnar;
  3. Left Tibial;
  4. Left Peroneal;
  5. Right Medial;
  6. Right Ulnar;
  7. Right Tibial;
  8. Right Peroneal
Number of patients with reduced/absent dCMAP amplitude at ≥1 site | up to 12 months
Number of patients with reduced/absent pCMAP amplitude at ≥1 site | up to 12 months
Proportion of patients with each score by each parameter of neurological examination | up to 12 months
Number of patients in the specific categories of the modified Rankin scale | up to 12 months
  1. Score 1 (no significant disability);
  2. Score 2 (slight disability);
  3. Score 3 (moderate disability);
  4. Score 4 (moderately severe disability);
  5. Score 5 (severe disability);
Proportion of patients with specific number of points according to Inflammatory Neuropathy Cause and Treatment (INCAT) upper extremity scale | up to 12 months
  1. 0 points;
  2. 1 point;
  3. 2 points;
  4. 3 points;
  5. 4 points;
  6. 5 points
Median number of points according to INCAT upper extremity scale | up to 12 months
Proportion of patients with specific number of points according to INCAT lower extremity scale | up to 12 months
  1. 0 points;
  2. 1 point;
  3. 2 points;
  4. 3 points;
  5. 4 points;
  6. 5 points
Median number of points according to INCAT lower extremity scale | up to 12 months
Mean and median number of points according to combined clinical and electrophysiological score | up to 12 months
To describe data on the results of genetic testing for ATTR in CTS patients undergoing surgery:Number and proportion of patients with specific TTR gene mutations | up to 12 months
  1. Val30Met;
  2. Ile107Val;
  3. Phe33Leu;
  4. Ala81Val;
  5. Ser23Asn;
  6. Ala25Thr;
  7. Val32Ala;
  8. Thr40Asn;
  9. Gly47Ala;
  10. Glu54Gln;
  11. Tyr69Phe;
  12. Glu92Lys;
  13. Thr119Met;
  14. Other
to assess general demographic and clinical characteristics of patients with ATTR PN in Russia - Proportion of patients with previously established incorrect diagnosis according to medical records, specifically with: | up to 12 months
  1. CIDP;
  2. Lumbar/sacral radiculopathy;
  3. Lumbar canal stenosis;
  4. Paraproteinaemic peripheral neuropathy;
  5. Chronic progressive sensory/sensorimotor axonal idiopathic PN;
  6. AL amyloidosis;
  7. Fibromyalgia;
  8. Other (specify);
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - proportion of patients with autonomic neurological manifestations, including specifically: | up to 12 months
  manifestations, including specifically:
  1. Orthostatic hypotension;
  2. Syncope;
  3. Gastrointestinal motility disorders - i. Constipation; ii. Early satiety; iii. Diarrhea; iv. Nausea, vomiting;
  4. Erectile dysfunction;
  5. Neurogenic bladder;
  6. Recurrent urinary infections;
  7. Anhidrosis;
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - proportion of patients with concomitant cardiac manifestations, including specifically: | up to 12 months
  1. Left ventricular hypertrophy;
  2. Left bundle branch block;
  3. Atrioventricular block;
  4. Heart failure with preserved ejection fraction;
  5. Elevated serum N-terminal-proB-type natriuretic peptide (NT-proBNP) concentration;
  6. Cardiac valve stenosis;
  7. Cardiac valve regurgitation;
  8. Tachyarrhythmia;
  9. Other (specify);
  10. None;
proportion of patients taking specific groups of cardiovascular medications at the time of CTS surgery and at the time of prospective visit: | up to 12 months
  1. Angiotensin converting enzyme inhibitor (ACEI) (specify);
  2. Angiotensin receptor blocker (ARB) (specify);
  3. Angiotensin receptor and neprilysin inhibitor (ARNI);
  4. Sodium-glucose transporter type 2 inhibitor (SGLT2i) (specify);
  5. Mineralocorticoid receptor antagonist (MRA) (specify);
  6. Beta-blocker (specify);
  7. Diuretic (specify);
  8. Other cardiovascular (CV) medications (specify);
  9. Other (specify);
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - proportion of patients with concomitant ophthalmologic manifestations, including specifically | up to 12 months
  1. Vitreous body inclusions (opacification);
  2. Glaucoma;
  3. Abnormal conjunctival vessels;
  4. Papillary abnormalities;
  5. Dry eye;
  6. Other (specify);
To describe data on the presence of cardiovascular, neurological and other comorbidities in Russian patients with ATTR PN - proportion of patients with concomitant musculoskeletal manifestations, including specifically: | up to 12 months
  1. Spinal stenosis;
  2. Osteoarthritis, including hip and knee arthroplasty;
  3. Trigger finger;
  4. Charcot's joints;
  5. Biceps tendon rupture;
  6. Rotator cuff injury;
  7. Other (specify);
proportion of patients with concomitant renal dysfunction, including specifically | up to 12 months
  1. Elevated SCr level (based on the local laboratory reference range);
  2. Decreased eGFR (<60 ml/min/1.73m2);
  3. Presence of albuminuria (≥30 mg/g creatinine (≥30 mg/g of creatinine or ≥30 mg/24h);
  4. Presence of proteinuria (according to urinalysis results);
  5. Ultrasound signs of amyloid nephropathy;
proportion of patients with confirmed length-dependent peripheral sensory-motor neuropathy based on NCS results | up to 12 months
proportion of patients with reduced peripheral sensory nerve conduction velocity at ≥1 site | up to 12 months
proportion of patients with reduced motor sensory nerve conduction velocity at ≥1 site | up to 12 months
proportion of patients with reduced/absent SAP amplitude at ≥1 site | up to 12 months
proportion of patients with reduced/absent dCMAP amplitude at ≥1 site | up to 12 months
proportion of patients with reduced/absent pCMAP amplitude at ≥1 site | up to 12 months
proportion of patients in the specific categories of the modified Rankin scale | up to 12 months
  -a) Score 1 (no significant disability); b) Score 2 (slight disability); c) Score 3 (moderate disability); d) Score 4 (moderately severe disability); e) Score 5 (severe disability
To assess general demographic characteristics of patients with ATTR PN in Russia - Mean age (years) at the primary CTS diagnosis | up to 12 months
To assess general demographic characteristics of patients with ATTR PN in Russia - Mean age (years) at the identification of bilateral involvement | up to 12 months
To assess general demographic characteristics of patients with ATTR PN in Russia - Mean age (years) at ATTR PN diagnosis | up to 12 months
To assess general demographic characteristics of patients with ATTR PN in Russia -Proportion of patients underwent CTS surgery (i.e. at least one surgery) | up to 12 months

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (13):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Ufa
  - Research Site, Yekaterinburg